CLINICAL TRIAL: NCT06240351
Title: A Pilot Study to Evaluate the Safety and Efficacy of Baricitinib in the Treatment of Frontal Fibrosing Alopecia (FFA)
Brief Title: A Study to Evaluate the Safety and Efficacy of Baricitinib in the Treatment of Frontal Fibrosing Alopecia (FFA)
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Boni Elewski, Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300009525; 2026154 (Other: Eli Lilly)
Record Dates: First submitted 2024-01-19; First posted 2024-02-05 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Frontal Fibrosing Alopecia
MeSH Terms: interventions — baricitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Baricitinib (Experimental): All patients will be treated with the active product, Baricitinib. Each patient will take 4mg of Baricitinib daily for 36 weeks.
  Interventions: Drug: Baricitinib 4 MG Oral Tablet

INTERVENTIONS:
Drug: Baricitinib 4 MG Oral Tablet — Baricitinib is a Janus kinase (JAK) inhibitor
  Other Names: Olumiant

SUMMARY:
The goal of this clinical trial is to evaluate the safety and efficacy of Baricitinib in the treatment of frontal fibrosing alopecia (FFA).

ELIGIBILITY:
Inclusion Criteria:

* Female at least 18 years of age, and able to provide informed consent
* Females who are post-menopausal defined, as not have menses for at least 12 months without an alternative medical cause and elevated follicle stimulating hormone in the postmenopausal range as measured during screening
* Have active FFA that has been diagnosed on or prior to screening visit.
* Have LPPAI score equal to or greater than 5 at screening.
* Have evidence of eyebrow loss at baseline
* Have evidence of hairline recession at baseline
* Have classic presentation with frontal loss of scalp hair
* Negative screening for tuberculosis (Quantiferon Gold, T-spot) within 3 months prior to screening or at the screening visit.
* Agree not to have a live vaccination during the study the exception is herpes zoster vaccine

Exclusion Criteria:

* Systemic treatments for FFA within 4 weeks of the baseline visit or 5 half lives whichever one is longer. (ex: finasteride, pioglitazone, hydroxychloroquine, or immunosuppressant medications, such as mycophenolate mofetil).
* Dutasteride within the last 6 months
* Have a LPPAI score less than 5 at screening
* Immunocompromised and with risk factors concerning to investigator for study participation
* Previous treatment with an oral JAK inhibitor
* Any condition in the opinion of the investigator which would interfere with the study assessments or procedure
* Subject is pregnant or breast feeding
* Surgical intervention including face lifts and micro-blading on the treatment areas
* Any intervention (facelifts micro blading) that could affect the treatment areas (i.e. scalp and eyebrows)
* Laser or phototherapy intervention on the treatment areas
* Have evidence of active TB or latent TB

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — This condition mostly impacts post-menopausal women.
Enrollment: 15 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
30% Change in Lichen Planopilaris Activity (LPPAI) Scores | From baseline to week 12, 24, and 36
  Percentage of patients achieving 30% change in LPPAI scores. LPPAI is a numeric scale that includes key signs and symptoms of FFA and allows for statistical comparison of disease activity. It captures patient reported symptoms (pruritus, pain, burning), clinical signs (erythema, perifollicular erythema, and scale), and other disease activity features (anagen pull and spreading). The total score distributes 30% weight to symptoms, 30% to signs, 25% to anagen pull, and 15% to spreading. The scale then ranges from 0-10 where 0 is no disease and 10 is worst disease.

SECONDARY OUTCOMES:
Improvement in Physician Global Assessment (PGA) | From baseline to week 12, 24, and 36
  Effectiveness of Baricitinib on improvement in Patient Global Assessment.This assessment is a scale from 0 to 4. 0 means clear skin while 4 means severe disease.
Change in inflammation on histology as seen on scalp biopsy | From baseline to week 12,24, and 36
  Effectiveness of Baricitinib on change of inflammation results on histology exam as seen on scalp biopsy. Degree of lymphocytic infiltrate will be assessed on biopsy and compared to cast thickness on trichoscopy (which correlates with severity of inflammatory changes on pathology).
Improvement in trichoscopic grading of peripheral cast by way of Tosti Scale | From baseline to week 12,24, and 36
  Effectiveness of Baricitinib on the improvement in trichoscopic grading of peripheral casts (scales). Degree of lymphocytic infiltrate will be assessed on biopsy and compared to cast thickness on trichoscopy by the Tosti Scale. This is a 3 grade measure with Grade 1 being minimum scaling while Grade 3 is maximum scaling.
Improvement in Eyebrow Assessment | From baseline to week 12,24, and 36
  Effectiveness of Baricitinib on the improvement of the eyebrow assessment. This is a survey for patients to answer. Answers range from 0 to 3. Answers of 0 mean "I have full eyebrows on each side" while answers of 3 mean " I have no or barely any eyebrow hairs.
Improvement in Visual Analog Scale (VAS) | From baseline to week 12,24, and 36
  Effectiveness of Baricitinib on the improvement of the Visual Analog Scale. This is a 10-point visual scale to rate whether the patient's FFA seems to be worse or resolved.

CONTACTS AND LOCATIONS:
Overall Officials: Boni Elewski, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States